CLINICAL TRIAL: NCT00559130
Title: Multi-Center, Efficacy Study of the MedaSorb CytoSorb™ Hemoperfusion Device as an Adjunctive Therapy in Subjects With Acute Respiratory Distress Syndrome (ARDS) or Acute Lung Injury (ALI) in the Setting of Sepsis
Brief Title: Efficacy Study of CytoSorb Hemoperfusion Device on IL-6 Removal in ARDS/ALI Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedaSorb Technologies, Inc (Industry)
Responsible Party: Dr. Robert Bartlett, MedaSorb Corp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-01
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; Sepsis
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury; Sepsis; Hemoperfusion
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CytoSorb Hemoperfusion — Daily hemoperfusion for 6 hours with CytoSorb device

SUMMARY:
The hypothesis of this study is use of CytoSorb hemoperfusion device as an adjunctive therapy to the standard of care in treating ARDS/ALI patients in the setting of sepsis will result in improved clearance of cytokines when compared to control patients receiving only the standard of care.

DETAILED DESCRIPTION:
Mortality rates from acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) range from 38.5 to 65%, with the lower mortality in acute lung injury than in ARDS.

ARDS/ALI is most often seen as part of a systemic inflammatory response syndrome (SIRS), particularly systemic sepsis. The lung findings parallel the damage in other tissues, namely, widespread destruction of the capillary endothelium, extravasation of protein rich fluid and interstitial edema. The alveolar basement membrane becomes damaged and fluid leaks into the airspaces, reducing lung compliance and causing ventilation-perfusion mismatch.

The most important causes of ALI/ARDS are sepsis, pneumonia, major trauma, pulmonary aspiration, near drowning, burns, inhalation of toxic gases (e.g. ammonia), fat embolism, amniotic fluid embolism, eclampsia, drug intoxication (e.g. aspirin), radiation injury and mechanical ventilation. Cox and colleagues have demonstrated in an ovine model of ARDS that there is intense acute inflammation in the trachea and bronchi from 3 to 48h after injury, with accumulation of neutrophils, fibrin and other plasma proteins, and mucus in airway lumens. Immunostaining for multiple cytokines (interleukin-8 (IL-8), IL-1beta, IL-1alpha, tumor necrosis factor-alpha (TNF-alpha), and vascular endothelial growth factor (VEGF)) are found in airway mucous glands, and the release of cytokines into the airway lumen are considered potentially highly significant in the progression of injury.

The importance of cytokines is being increasingly realized in mechanical lung injury (a common cause of ALI/ARDS) associated with mechanical ventilation (MV). Here the pathway is identical with release of cytokines/chemokines which potentiate the extravasation, activation, and recruitment of leukocytes, causing ventilator-associated lung injury (VALI) and ventilator-induced lung injury (VILI). Moreover, VALI/VILI can perpetuate the chronic inflammatory response during ALI/ARDS and multiple organ dysfunction syndrome (MODS).

The purpose of this study is to evaluate the reduction of cytokines, using the CytoSorb device, on primary and secondary endpoints

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent document (ICD)
* Male or female ≥ 18 and ≤ 80 years of age.
* Subjects must have diagnosis of ARDS or ALI, based on ARDSNet Definition, established within last 72 hours, confirmed by clinical, radiological, or physiologic findings
* Subject must be intubated
* ≤ 3 days on a ventilator prior to enrollment
* Subjects must have confirmed diagnosis of sepsis
* Subject must have had at least 24 hours of antibiotic therapy
* Pre-menopausal female subjects must have negative pregnancy test.
* Subject must be available for periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study. Subject must have permanent home address to allow completion of 60 day follow-up.
* Subject or health care proxy has the ability to understand and willingness to sign the informed consent form.

Exclusion Criteria:

* Currently participating in another clinical study involving investigational chemical compound, biologic, or device within the last 30 days prior to the start of this trial.
* Neuromuscular disease that impairs the ability to ventilate spontaneously, such as C5 or higher spinal cord injury, amyotrophic lateral sclerosis, Guillain-Barré syndrome and myasthenia gravis.
* Increased intracranial pressure, tricyclic antidepressant overdose, hemoglobin SS, hemoglobin SC or other conditions where hypercapnia would be contraindicated.
* Severe chronic respiratory disease including hospitalization within last 6 months for respiratory failure.
* Morbid obesity (Body Mass Index ≥40 kg/m2).
* Burns > 30% BSA, bone marrow transplant, lung transplant or end stage hepatic liver failure.
* Subject with mean arterial pressure ≤ 60 mmHg regardless of use of pressor agents.
* Subject with active malignancy receiving chemotherapy or radiation treatment within last 60 days.
* Subjects with AIDS, CD4 count of < 200 or 14%, or the presence of an AIDS defining illness (HIV+ subjects may be enrolled)
* Subject with acute coronary syndrome.
* Subjects with decompensated heart failure with New York Heart Association (NYHA) classification IV
* Subjects with Chronic Kidney Disease (CKD) stage 5 will be excluded
* Subjects with end stage hepatic liver failure
* Subjects on immunosuppressive agents, excluding corticosteroids
* Platelets ≤ 20,000/mm3
* Subjects on anti-TNF therapy
* Subjects about to receive or receiving drotrecogin alpha (Xigris) therapy
* Subject is pregnant or breastfeeding.
* Subject has a known allergy to any component of the CytoSorb hemoperfusion device
* Subject has any active disease condition that could limit compliance with the study procedure, including but not limited to the following: acute coronary syndrome, life-threatening cardiac arrhythmia, or psychiatric or social conditions, considered by investigator(s) to preclude successful completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Relative IL-6 levels as a percent (%) of baseline will be lower in subjects receiving CytoSorb treatment in conjunction with the standard of care as compared to control subjects receiving only the standard of care for ARDS/ALI in the setting of sepsis. | 7 Days

SECONDARY OUTCOMES:
Ventilator Free Days, Reduction cytokines TNF-α, IL-1b, IL-10, CRP, 28-day all cause mortality, Oxygen Index (OI), P/F ratios, MODS scores | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Kuhlmann, Prof. Dr., Principal Investigator — Vivantes Klinikum
Locations (6):
- Germany (6):
  - Aachen
  - Berlin
  - Bonn
  - Erfurt
  - Göttingen
  - Kiel